CLINICAL TRIAL: NCT01904786
Title: Melatonin Treatment for Newborn Infants With Moderate to Severe Hypoxic Ischemic Encephalopathy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment of suitable candidates
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLU22484
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-01

CONDITIONS: Newborn Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic Ischemic Encephalopathy; Newborn; Outcomes; Melatonin
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): Melatonin 40 mg every 8 hours for a total of six doses given over 48 hours orally (per nasogastric tube).
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo consists of the solvent solution without melatonin. Solvent solution consists of 5 mL of saline/alcohol mixture in a ratio of 90:1
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Melatonin
  Arms: Melatonin
Drug: placebo
  Arms: Placebo

SUMMARY:
During the birth process certain conditions can cause oxygen delivery and/or blood flow to the baby's brain to become interrupted. This can cause permanent brain damage. Brain damage occurs in two phases. The first occurs at the time of injury when brain cells in the affected area 'die'. There is nothing that can be done about this. The second phase of injury occurs over the next few days. This second phase is caused by inflammation and release of toxic chemicals from the injured site. Cooling the baby to a temperature of 92.5° F, for 3 days has been shown to reduce the second phase of injury and bran death. All babies will receive the benefit of cooling. Although cooling helps it does not completely stop the second phase of injury.

Melatonin is a naturally occurring hormone that is produced by the brain, and helps regulate the sleep-wake cycle. It has the potential to stop the second phase of brain injury by inhibiting inflammation and release of toxic chemicals. The reason for this research is to find out if melatonin can or cannot improve the outcome of babies with this kind of brain damage. Every baby enrolled in the study has a 50:50 chance of getting melatonin. A total of six doses of medicine will be given. The baby's brain function will be assessed by an EEG, brain oxygen monitoring, and a neurologic examination at 18 months of life. All of these are routinely used as part of standard care for patients with this kind of problem. The only difference is that half the babies enrolled in the study will get the drug called melatonin and the other half will receive placebo. The dose of melatonin being used in the study is higher than the amount normally produced by the body. No side-effects of this dose have been reported in other research studies using melatonin in newborn and premature babies.

DETAILED DESCRIPTION:
This is a double-blind randomized study. All babies less than eight hours old, admitted to the NICU at Cardinal Glennon Children's Medical Center, with moderate to severe HIE that qualify for whole body cooling will be eligible for enrollment in the study. Whole body cooling is part of standard treatment for babies with moderate to severe HIE, and the criteria for diagnosis and cooling are well established. After consent is obtained babies will be randomly assigned to melatonin treatment or control groups (standard treatment) using a 4-block randomization design, by opening a sealed opaque sequentially numbered envelope by the study pharmacist. A log of assignments will be maintained by the study pharmacist. The clinical team will be blinded as to the assignment. Patients assigned to melatonin treatment will receive 40 mg melatonin (PureBulk, CA, USA) in 5 mL of vehicle (1:90 mix ethanol/saline) every 8 hours for a total of six doses. Patients assigned to the control group will receive 5 mL of vehicle only every 8 hours for a total of six doses. All doses will be administered via a nasogastric tube by the nurse assigned to the patient. Placement of a nasogastric tube is part of standard care for babies with HIE. Administration of the first dose within eight hours of life is mandatory for the study.

EEG analysis is part of standard neurologic evaluation for patients with HIE, and is done once the patient has been rewarmed to normal body temperature (by 78-80 hours after starting whole body cooling). A 24 hour multichannel video-EEG (Nihon Kohden 9100A, Nihon Kohden USA Inc.) using the 10-20 system of electrode placement modified for neonates will be performed between 80 and 100 hours after initiation of the cooling protocol. The duration of each seizure will be added together for the entirety of the recording to obtain the seizure burden (total seizure time).

Anticonvulsant treatment will assessed at the time of discharge whether the patient is on any, one, or more anticonvulsants.

Cerebral tissue oxygenation (rSO2) will be monitored non-invasively by applying the NIRS probe to the forehead and attaching it to the INVOS monitor (Somanetics, MI, USA). The probe is very similar to the oxygen saturation oximeter probe that is routinely used in newborns. Cerebral tissue oxygenation will be continuously monitored until re-warming is complete. Data will be collected at the start of monitoring and then every six hours.

A brain MRI is not required for the study, but if it is obtained then the results may be included in the data collected.

ELIGIBILITY:
Inclusion Criteria:

* Infants with moderate to severe hypoxic ischemic encephalopathy ≥36 weeks
* First dose of study drug given within 8 hours of birth

Exclusion Criteria:

* Major chromosomal or congenital defects

Ages: 1 Hour to 8 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopment at 18 months of life (BSID-III) | 18 months
  The Bayley Scales of Infant Development III exam will be administered at 18 months of life to assess neurodevelopment.

SECONDARY OUTCOMES:
Seizure burden | Assessed on day 3-4 of life
Reduction in Burst Suppression | Assessed on day 3-4 of life
Improved cerebral oxygenation | First 3-4 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Sadiq, MD, Principal Investigator — St. Louis University
Locations (1):
- Cardinal Glennnon Children's Medical Center, St Louis, Missouri, United States